CLINICAL TRIAL: NCT06782841
Title: The Effects of GMA-TULIP, I-gel, and BlockBuster Laryngeal Mask in Surgeries With Lateral Position Under General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.134
Record Dates: First submitted 2025-01-05; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-07

CONDITIONS: Oropharyngeal Leak Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GMA-TULIP Laryngeal Mask Group（D1 Group） (Experimental): After the anesthesia induction, use the GMA-TULIP laryngeal mask as the airway ventilation device.
  Interventions: Device: GMA-TULIP Laryngeal Mask
- i-gel Laryngeal Mask Group（D2 Group） (Active Comparator): After the anesthesia induction, use the i-gel laryngeal mask as an airway ventilation device.
  Interventions: Device: i-gel Laryngeal Mask
- BlockBuster Laryngeal Mask Group（D3 Group） (Active Comparator): After the anesthesia induction is over, use the BlockBuster laryngeal mask as the airway ventilation device.
  Interventions: Device: BlockBuster Laryngeal Mask

INTERVENTIONS:
Device: GMA-TULIP Laryngeal Mask — After the anesthesia induction, use the GMA-TULIP laryngeal mask as the airway ventilation device.
  Arms: GMA-TULIP Laryngeal Mask Group（D1 Group）
Device: i-gel Laryngeal Mask — After the anesthesia induction, use the i-gel laryngeal mask as an airway ventilation device.
  Arms: i-gel Laryngeal Mask Group（D2 Group）
Device: BlockBuster Laryngeal Mask — After the anesthesia induction is over, use the BlockBuster laryngeal mask as the airway ventilation device.
  Arms: BlockBuster Laryngeal Mask Group（D3 Group）

SUMMARY:
To compare the efficacy and safety of traditional inflatable laryngeal mask, i-gel non-inflatable laryngeal mask and GMA-TULIP non-inflatable laryngeal mask in surgeries with lateral position under general anesthesia, so that providing evidence for the selection of laryngeal mask in surgeries with lateral position.

DETAILED DESCRIPTION:
Laryngeal mask and tracheal intubation are the two most commonly used airway management methods for patients under general anesthesia. Compared with tracheal intubation, laryngeal mask is only placed in the throat without the need for laryngoscope to expose the glottis, not entering the glottis and trachea, so it will not cause mechanical damage to the vocal cords and trachea. Moreover, the insertion of laryngeal mask reduces the excitation of sympathetic and vagus nerves, has a relatively mild effect on physiological status, and significantly reduces cardiovascular reactions, which is convenient for maintaining hemodynamic stability during anesthesia induction and patients can tolerate the tube better without coughing or agitation during recovery from the anesthesia. Therefore, laryngeal masks are currently widely used in airway management during general anesthesia. Studies have shown that about 3 million patients in the UK National Health Service system receive anesthesia surgery with different types of airway management every year, and the use of laryngeal masks is higher than that of tracheal intubation, accounting for about 56.2%.

Since its introduction, many new laryngeal masks have been improved and applied to clinical practice based on the classic laryngeal mask. A key indicator for evaluating the performance of laryngeal masks is their sealing effect on the airway. Currently, laryngeal masks are mainly divided into two categories: inflatable laryngeal masks and non-inflatable laryngeal masks. Inflatable laryngeal masks are traditional types, including BlockBuster, Superme, ProSeal, and Fastrach, which are the most widely used in clinical practice. Non-inflatable laryngeal masks are designed with a mirror image of the throat opening and use thermoplastic elastomer materials to achieve a gas tightness effect similar to that of inflatable laryngeal masks. The i-gel laryngeal mask is currently the most commonly used non-inflatable type. A meta-analysis found that the sealing pressure of the i-gel laryngeal mask is higher than that of traditional inflatable laryngeal masks, indicating better airway sealing performance for non-inflatable laryngeal masks. The GMA-TULIP non-inflatable laryngeal mask is a new type of non-inflatable laryngeal mask with advantages such as a C-shaped double gastric tube channel, a stable platform for the tongue base, a soft tissue sealing ring, a prominent epiglottis attachment, and a design that matches the anatomical structure of the throat opening. Compared with inflatable laryngeal masks, the GMA-TULIP mask is more in line with anatomical positioning design, theoretically providing higher sealing effect on the airway.

Although the laryngeal mask has been successfully applied to the airway management of surgeries with lateral position under general anesthesia, its widespread use is limited due to the special position of lateral position, which may lead to laryngeal mask displacement, poor airway tightness, and air leakage. Therefore, exploring a laryngeal mask with better airway sealing effect in surgeries with lateral position under general anesthesia will help promote the clinical application of laryngeal mask, reduce airway injury and hemodynamic fluctuation, and improve patient comfort. To this end, this project plans to compare the application effects of traditional inflatable BlockBuster laryngeal mask, i-gel non-inflatable laryngeal mask, and GMA-TULIP non-inflatable laryngeal mask in surgeries with lateral position under general anesthesia, providing clinical evidence for the selection of laryngeal mask in surgeries with lateral position under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients received surgeries in lateral position with an estimated surgery duration of less than 3 hours under general anesthesia.
2. Ages between 18 to 80, and body mass index less than 28 kg/m².
3. American Society of Anesthesiologists (ASA) Grades I-III.
4. Patients are willing to participate and be able to understand and sign an informed consent form.

Exclusion Criteria:

1. Individuals with an open bite of less than 2cm.
2. Individuals with a history of obvious regurgitation of gastric contents and risk factors for aspiration.
3. Patients with combined pharyngeal and laryngeal lesions.
4. Predicting difficult airway patients.
5. Hearing, intellectual, communication, and cognitive impairments.
6. Any reason that prevents cooperation with the study or that the researcher deems inappropriate for inclusion in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
oropharyngeal leak pressure | 1 minute after the laryngeal mask is successful inserted, 5 and 30 minutes after the lateral position
  After the laryngeal mask is successful inserted, set the fresh gas flow to 3 L/min in manual mode, turn the APL valve to 30 cmH2O, then listen to the neck. When hearing the sound of air leakage, the peak airway pressure at this time is the oropharyngeal leak pressure.

SECONDARY OUTCOMES:
The rate of first-insertion success | 1 minute after the first-attempt insertion of the laryngeal mask
  The successful insertion is defined as oropharyngeal leak pressure higher than 20 cmH2O and grade 1-2 of the laryngeal view under the fibreoptic bronchoscopy (indicating the accuracy of laryngeal mask positioning).
The rate of total-insertion success | 1 minute after the airway is successfully controlled.
  The total successful insertion is defined as ventilation with the allocated laryngeal mask after anesthesia induction
Time of insertion | 1 minute after successful insertion of the laryngeal mask
  Insertion time was defined as the time from the opening of the mouth by the operator to the positively insert the laryngeal mask. The time of glottic examination, adjustment between two ventilation insertions, and ventilation was not measured as ventilation insertion time.
Times of laryngeal mask adjustment before the successful insertion | 1 minute after the airway is successfully controlled.
  The times of laryngeal mask adjustments before successful laryngeal mask insertion.
Success rate of gastric tube insertion through laryngeal mask | 1 minute after the laryngeal mask is successful inserted
  After the laryngeal mask is successful inserted, a fully lubricated 14F gastric tube was inserted through its esophageal drainage tube
Airway plateau pressure | 1 minute after the laryngeal mask is successful inserted, 5 and 30 minutes after the lateral position
  Plateau airway pressure refers to the pressure that a certain amount of gas remains in the lungs against the entire closed system at the end of the passage of air, before the beginning of exhalation. Airway plateau pressure was measured by the anesthesia machine automatically.
Peak airway pressure | 1 minute after the laryngeal mask is successful inserted, 5 and 30 minutes after the lateral position
  Peak pressure refers to the maximum pressure produced by the airflow in the closed circuit each time the ventilator delivers a certain amount of gas from the endotracheal tube to the patient's lungs. Peak airway pressure was measured by the anesthesia machine automatically.
grade of view on fibreoptic bronchoscopy (indicating the accuracy of laryngeal mask positioning) | 1 minute after the laryngeal mask is successful inserted, 5 and 30 minutes after the lateral position
  After successful insertion of the laryngeal mask, fiberoptic bronchoscopy was used and graded according to the degree of glottic and epiglottis exposure by a 4-point scale system: 1, full view of glottis; 2, vocal cords, arytenoids, and inferior surface of epiglottis visible; 3, only superior surface of epiglottis visible; 4, no part of epiglottis or larynx visible. The grades 1 and 2 were defined as optimal fiberscopic view.
Times of laryngeal mask adjustment during the operation | From 1 minute after the beginning of anesthesia to 1 minute after the end of anesthesia
  the times of the laryngeal mask adjustment during the operation were recorded
Times of intraoperative air leakage | From 1 minute after the beginning of anesthesia to 1 minute after the end of anesthesia
  intraoperative air leakage is defined as hearing the sound of air leakage at the neck during the operation
Active mouth bleeding rate | 1 minute after laryngeal mask removal
  After the laryngeal mask was removed, record whether active bleeding occurred at the patient's mouth
incidence of blood staining on the laryngeal mask | 1 minute after the laryngeal mask was withdrawn
  When the laryngeal mask was pulled out, the laryngeal mask was stained with blood
The incidence of regurgitation | From 1 minute after the beginning of anesthesia to 1 minute after the end of anesthesia
  The regurgitation is defined as seeing the gastric content in the mouth
The incidence of aspiration | From 1 minute after the beginning of anesthesia to 1 minute after the end of anesthesia
  The aspiration is defined as seeing the gastric content in the trachea
The incidence of cough | From 5 minutes before to 5 minutes after the laryngeal mask withdrawal.
  When the laryngeal mask was pulled out, record whether the patient has cough or not.
Severity of sore throat | 10 minutes, 2 hours, 24 hours, 48 hours, and 72 hours after surgery
  The Prince-Henry score was used to evaluate the degree of sore throat: 0, no pain when coughing; 1, pain only when coughing; 2, pain when breathing deeply, but not at rest; 3, pain at rest, but mild and tolerable; 4, excruciating pain at rest, respectively.
Length of surgery | 1 minute after the end of surgery
  The end of the surgery time minus the start of the surgery time
Time of laryngeal mask application | 1 minute after the laryngeal mask is withdrawn
  The time of laryngeal mask withdrawn minus the time of successful laryngeal mask insertion is the time of laryngeal mask application
The incidence of hoarseness | 10 minutes, 2 hours, 24 hours, 48 hours, and 72 hours after surgery
  Record whether the patient is hoarse when speaking
The incidence of dysphagia | 10 minutes, 2 hours, 24 hours, 48 hours, and 72 hours after surgery
  Check the patient can swallow or not
Heart rate | 1 minute before laryngeal mask insertion or withdrawn, and 1 minute after the laryngeal mask is inserted or withdrawn
  Heart rate
systolic blood pressure | 1 minute before laryngeal mask insertion or withdrawn, and 1 minute after the laryngeal mask is inserted or withdrawn
  systolic blood pressure
diastolic blood pressure | 1 minute before laryngeal mask insertion or withdrawn, and 1 minute after the laryngeal mask is inserted or withdrawn
  diastolic blood pressure
mean arterial pressure | 1 minute before laryngeal mask insertion or withdrawn, and 1 minute after the laryngeal mask is inserted or withdrawn
  mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Bing Chen, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available with the responding author when required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available when publish and keep it for 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal.